CLINICAL TRIAL: NCT01796925
Title: Clinical Study of the aura6000™ Targeted Hypoglossal Implantable Neurostimulation (THN) Sleep Therapy System
Brief Title: Targeted Hypoglossal Neurostimulation Study #2
Acronym: THN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ImThera Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: LivaNova (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMT2012-02
Record Dates: First submitted 2013-02-14; First posted 2013-02-22 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiration Disorders; Signs and Symptoms, Respiratory; Syndrome, Obstructive Sleep Apnea
Keywords: Apnea; Respiration Disorders; Signs and Symptoms; Signs and Symptoms, Respiratory; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiratory Tract Diseases; Sleep Disorders, Intrinsic; Sleep Disorders; Nervous System Diseases
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiration Disorders; Signs and Symptoms, Respiratory; Apnea; Signs and Symptoms; Respiratory Tract Diseases; Sleep Disorders, Intrinsic; Sleep Wake Disorders; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aura6000 THN Therapy (Experimental): The aura6000 THN system will be implanted and activated for nightly therapy during sleep.
  Interventions: Device: aura6000 THN System

INTERVENTIONS:
Device: aura6000 THN System — The aura6000 device is an implanted hypoglossal nerve stimulator designed to maintain wakeful muscle tone of the tongue during sleep. It is implanted through a short surgical procedure. The implant is programmed to provide the optimal stimulation parameters for the patient. The therapy is controlled by a hand-held remote control allowing the patient to start, stop, and pause the therapy during times of sleep.

SUMMARY:
The objective of the study is to confirm the safety and efficacy in patients utilizing the aura6000 System for the treatment of Obstructive Sleep Apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* AHI >20
* Noncompliant to CPAP
* Willing to provide informed consent
* Willing to comply with all follow-up visits and evaluations

Exclusion Criteria:

* BMI limits
* COPD
* Central Sleep Apnea
* Anatomic variations interfering with device placement or stability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Reduction in Apnea-Hypopnea Index (AHI) | 3, 6, and 12 months post implant
  Change from baseline in AHI measured through in-lab polysomnography (PSG).
Reduction in Oxygen Desaturation Index (ODI) | 3, 6, and 12 months post implant
  Change from baseline in ODI measured through in-lab polysomnography (PSG).
Freedom from Serious Adverse Events (SAE) | 1 and 12 months post implant
  Adverse events and Serious Adverse events post-operatively

SECONDARY OUTCOMES:
Improvement in sleep fragmentation | 3, 6, and 12 months post-implant
  Mean change in microarousal index as compared to baseline.
Improvement in SAQLI | 3, 6, and 12 months post implant
  Mean change in SAQLI (Sleep Apnea Quality of Life Index) as compared to baseline.
Improvement in ESS | 3, 6, and 12 months post implant
  Mean change in ESS (Epworth Sleepiness Scale) as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rodenstein, MD, PhD, Principal Investigator — Clinique Univ. Saint-Luc; Ofer Jacobowitz, MD PhD, Principal Investigator — Hudson Valley ENT
Locations (9):
- United States (4):
  - Sharp Rees Stealy Medical Center, San Diego, California
  - Porter Adventist Hospital, Denver, Colorado
  - Chicago ENT, Chicago, Illinois
  - Orange Regional Medical Center, Middletown, New York
- Clinique Univ. Saint-Luc, Brussels, Belgium
- Pitié-Salpêtrière Hospital, Paris, France
- Germany (2):
  - Advanced Sleep Research, Berlin
  - St. Joseph-Stift, Bremen
- G.B. Morgagni- L. Pierantoni Hospital, Forlì, Italy

REFERENCES:
- [Background] Zaidi FN, Meadows P, Jacobowitz O, Davidson TM. Tongue anatomy and physiology, the scientific basis for a novel targeted neurostimulation system designed for the treatment of obstructive sleep apnea. Neuromodulation. 2013 Jul-Aug;16(4):376-86; discussion 386. doi: 10.1111/j.1525-1403.2012.00514.x. Epub 2012 Aug 31. PMID 22938390
- [Background] Mwenge GB, Rombaux P, Dury M, Lengele B, Rodenstein D. Targeted hypoglossal neurostimulation for obstructive sleep apnoea: a 1-year pilot study. Eur Respir J. 2013 Feb;41(2):360-7. doi: 10.1183/09031936.00042412. Epub 2012 May 17. PMID 22599356